CLINICAL TRIAL: NCT01688440
Title: "ETCare": A Phase II, Safety and Preliminary Efficacy Trial
Brief Title: ETCare: Safety and Preliminary Efficacy Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Principal Investigator, Robert D. Christensen, MD, Director, Neonatology Research, Intermountain Health Care, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05.018
Record Dates: First submitted 2008-05-12; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Endotracheal Cares; Neonate; TAC's; Endotracheal Suctioning; Tracheal Aspirate Culture; Oral Cares; Neonate oxygen Therapy
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- #1 Respiratory Care Solution (Experimental): Low sodium physiologically based airway care solution.
  Interventions: Other: #1 Respiratory Care Solution

INTERVENTIONS:
Other: #1 Respiratory Care Solution — Respiratory care solution.

SUMMARY:
When babies are sick, or are born prematurely, they sometimes need an endotracheal (ET) tube to assist their breathing and/or a nasal canula. The investigators must periodically irrigate the ET tube to prevent them from being plugged up by secretions. The investigators also, due to the drying effects of nasal canula, periodically moisten the nasal passages of babies. Presently 0.9% saline is the solution being used for moistening of the ET tube, nose, as well as oral cares will infant is not eating. However, scientists have recently learned that saline can destroy the body's natural antibacterial properties in the windpipe, nose, and mouth.

The investigators have developed a new solution to be used in place of saline for endotracheal (ET), nasal, and oral cares. The investigators' new solution is patterned after the natural fluid in the windpipe, nose, and mouth.

Study Hypothesis:

1. Patients who receive ETCare will have no increase in adverse events related to its administration, compared with 0.9% saline.
2. Patients who receive ETCare will have a lower proportion of tracheal aspirates where pathogens are reported.
3. Patients who receive ETCare will have a lower proportion of tracheal aspirates where leukocytes are reported.
4. Patients who receive ETCare will have fewer (risk-adjusted) days of supplemental oxygen.

DETAILED DESCRIPTION:
Normal saline (0.9% sodium chloride) is used by virtually all neonatal intensive care units to periodically irrigate the endotracheal tube of neonates who require mechanical ventilation. This practice is intended to reduce the risk that thick secretions will occlude the endotracheal tube. Normal saline is also occasionally used to periodically clear the nasal passages of neonates on nasal CPAP or nasal canula oxygen. It is also occasionally used as a means of periodically moistening the mouth of neonates who have an endotracheal tube in place, because the tube prevents lip apposition and results in a dry mouth.

The problem with the current method of using normal saline for periodic endotracheal, nasal, and/or oral care is that high concentrations of sodium and chloride have recently been found to rapidly and completely inactivate the natural antimicrobial properties of tracheal effluent, nasal secretions, and saliva. Tracheal secretions, nasal secretions, and saliva contain potent antibacterial substances. One such that was recently described is a 37 amino acid peptide with widespread antimicrobial properties, termed "LL-37". It has recently been shown that 0.9% saline inactivates the antimicrobial properties of LL-37 and significantly damages the overall antibacterial actions of tracheal secretions, nasal secretions, and saliva. Further research has shown that the high sodium and chloride content of saliva of patients with cystic fibrosis inactivates the antimicrobial properties, thus partly explaining the high incidence of airway infections in these patients. Moreover, a family with deficient LL-37 has been described in Sweden, and these individual all have chronic gingivostomatitis and airway infections. Therefore, our current practice of instilling 0.9% sodium chloride likely inactivates the major innate anti-microbial defense system of the upper airway. Perhaps reducing immune capacity in the upper airway with this practice unwittingly contributes to the high incidence of upper airway infections among intubated neonates.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient in the NICU of either McKay-Dee Hospital or LDS Hospital.
* Be <24 hrs old at the time of study entry.
* Have an endotracheal tube in place.
* Be expected, by declaration of the attending neonatologist, to have an endotracheal tube for at least the next 48 hrs.
* Have the informed consent document signed by the parent or responsible guardian

Exclusion Criteria:

* They have what the attending neonatologist judges to be a "lethal" congenital abnormality.
* They have a condition that is likely (by judgment of the attending neonatologist) to require transfer to Primary Children's Medical Center before the endotracheal tube has been electively removed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events related to administration. | To discharge home (about one month).
  Renal hematological and hepatic function.

SECONDARY OUTCOMES:
Feasibility and immediate intolerance | Day of administration (one day)
  Desaturation, bradycardia, tachydardia, hypotension, or hypertension or skin rashes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Christensen, MD, Principal Investigator — Interountain Healthcare
Locations (2):
- United States (2):
  - McKay-Dee Hospital Center, Ogden, Utah
  - LDS Hospital Center, Salt Lake City, Utah